CLINICAL TRIAL: NCT06697730
Title: Study of the Incidence and Prognosis of Intrahospital Acute Kidney Injury
Acronym: SIPARIO-1
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 5261_1
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; hospitalized
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized Patients: All patients hospitalized from 01/01/2019 to 12/31/2023.

SUMMARY:
The goal of this observational study is to investigate the epidemiology of acute kidney injury in hospitalized patients. The main question it aims to answer is: how frequent is the development of acute kidney injury in patients who are hospitalized? Data from participants will be retrospectively collected from medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised from 01/01/2019 to 31/12/2023
* Availability of a Hospital Discharge Form
* At least one serum creatinine (sCr) determination available

Exclusion Criteria:

* Day-hospital admission
* Discharge after an emergency room admission without hospital admission
* Stage IV and V CKD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all patients admitted to the reference hospital during the indicated time frame; in particular, all patients for whom sufficient data are available to establish the presence or absence of a diagnosis of AKI will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 43000 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of intra-hospital Acute Kidney Injury | From 01/01/2019 to 12/31/2023

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury in different hospital wards | From 01/01/2019 to 12/31/2023
Association between Acute Kidney Injury development and major discharge diagnoses | From 01/01/2019 to 12/31/2023
Rate of re-hospitalisation in Acute Kidney Injury (AKI) and non-AKI patients | From 01/01/2019 to 12/31/2023
Intra-hospital mortality rate in patients who developed AKI compared to those who did not | From 01/01/2019 to 12/31/2023
Incidence of AKI associated with thrombotic microangiopathy | From 01/01/2019 to 12/31/2023
  Comparison between hospital discharge forms and presumptive diagnosis formulated by parametric algorithms based on haematochemical tests performed during hospitalisation

IPD SHARING:
Plan to Share IPD: Undecided